CLINICAL TRIAL: NCT01431287
Title: A Randomised, Double-blind, Parallel Group Study to Assess the Efficacy and Safety of 52 Weeks of Once Daily Treatment of Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination (2.5 µg / 5 µg; 5 µg / 5 µg) (Delivered by the Respimat® Inhaler) Compared With the Individual Components (2.5 µg and 5 µg Tiotropium, 5 µg Olodaterol) (Delivered by the Respimat® Inhaler) in Patients With Chronic Obstructive Pulmonary Disease (COPD) [TOnado TM 2]
Brief Title: Tiotropium +Olodaterol Fixed Dose Combination (FDC) Versus Tiotropium and Olodaterol in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.6; 2009-010669-22 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-09-08; First posted 2011-09-09 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; Tiotropium Bromide; olodaterol

ARMS (5):
- tiotropium+olodaterol high dose FDC (Experimental): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium + olodaterol; Device: Respimat
- tiotropium+olodaterol low dose FDC (Experimental): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium + olodaterol; Device: Respimat
- olodaterol (Active Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: olodaterol; Device: Respimat
- tiotropium low dose (Active Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium; Device: Respimat
- tiotropium high dose (Active Comparator): Once daily 2 puffs solution for inhalation Respimat
  Interventions: Drug: tiotropium; Device: Respimat

INTERVENTIONS:
Drug: tiotropium + olodaterol — fixed dose combination
  Arms: tiotropium+olodaterol low dose FDC
Drug: tiotropium + olodaterol — fixed dose combination
  Arms: tiotropium+olodaterol high dose FDC
Drug: tiotropium — low dose or high dose
  Arms: tiotropium low dose
Drug: tiotropium — low dose or high dose
  Arms: tiotropium high dose
Drug: olodaterol — one dose only
  Arms: olodaterol
Device: Respimat — Respimat inhaler

SUMMARY:
The overall objective of this study is to assess the efficacy and safety of 52 weeks once daily treatment with orally inhaled tiotropium + olodaterol FDC (delivered by the RESPIMAT Inhaler) compared with the individual components (tiotropium, olodaterol) (delivered by the RESPIMAT Inhaler) in patients with COPD.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of chronic obstructive pulmonary disease.
2. Relatively stable airway obstruction with post FEV1< 80% predicted normal and post FEV1/FVC <70%.
3. Male or female patients, 40 years of age or older.
4. Smoking history of more than 10 pack years.

Exclusion criteria:

1. Significant disease other than COPD
2. Clinically relevant abnormal lab values.
3. History of asthma.
4. Diagnosis of thyrotoxicosis
5. Diagnosis of paroxysmal tachycardia
6. History of myocardial infarction within 1 year of screening visit
7. Unstable or life-threatening cardiac arrhythmia.
8. Hospitalization for heart failure within the past year.
9. Known active tuberculosis.
10. Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years
11. History of life-threatening pulmonary obstruction.
12. History of cystic fibrosis.
13. Clinically evident bronchiectasis.
14. History of significant alcohol or drug abuse.
15. Thoracotomy with pulmonary resection
16. Oral ß-adrenergics.
17. Oral corticosteroid medication at unstable doses
18. Regular use of daytime oxygen therapy for more than one hour per day
19. Pulmonary rehabilitation program in the six weeks prior to the screening visit
20. Investigational drug within one month or six half lives (whichever is greater) prior to screening visit
21. Known hypersensitivity to ß-adrenergic drugs, anticholinergics, BAC, EDTA
22. Pregnant or nursing women.
23. Women of childbearing potential not using a highly effective method of birth control
24. Patients who are unable to comply with pulmonary medication restrictions

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2539 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (240):
- United States (38):
  - 1237.6.01106 Boehringer Ingelheim Investigational Site, Greer, California
  - 1237.6.01120 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1237.6.01131 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 1237.6.01117 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1237.6.01118 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1237.6.01126 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1237.6.01109 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1237.6.01134 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1237.6.01107 Boehringer Ingelheim Investigational Site, Couer d'Alene, Idaho
  - 1237.6.01110 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1237.6.01128 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1237.6.01130 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1237.6.01104 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1237.6.01116 Boehringer Ingelheim Investigational Site, Plymouth, Minnesota
  - 1237.6.01121 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1237.6.01123 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1237.6.01129 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1237.6.01136 Boehringer Ingelheim Investigational Site, Marlton, New Jersey
  - 1237.6.01108 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1237.6.01127 Boehringer Ingelheim Investigational Site, Bayside, New York
  - 1237.6.01139 Boehringer Ingelheim Investigational Site, Great Neck, New York
  - 1237.6.01135 Boehringer Ingelheim Investigational Site, Charlotte, North Carolina
  - 1237.6.01114 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1237.6.01102 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1237.6.01115 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1237.6.01101 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1237.6.01113 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1237.6.01122 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1237.6.01132 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1237.6.01137 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1237.6.01111 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.6.01105 Boehringer Ingelheim Investigational Site, Union, South Carolina
  - 1237.6.01138 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1237.6.01124 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 1237.6.01112 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1237.6.01133 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1237.6.01125 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1237.6.01103 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Austria (6):
  - 1237.6.43006 Boehringer Ingelheim Investigational Site, Feldbach
  - 1237.6.43005 Boehringer Ingelheim Investigational Site, Gänserndorf
  - 1237.6.43002 Boehringer Ingelheim Investigational Site, Innsbruck
  - 1237.6.43004 Boehringer Ingelheim Investigational Site, Leoben
  - 1237.6.43001 Boehringer Ingelheim Investigational Site, Linz
  - 1237.6.43003 Boehringer Ingelheim Investigational Site, Salzburg
- Belgium (9):
  - 1237.6.32005 Boehringer Ingelheim Investigational Site, Brussels
  - 1237.6.32007 Boehringer Ingelheim Investigational Site, Brussels
  - 1237.6.32004 Boehringer Ingelheim Investigational Site, Ghent
  - 1237.6.32002 Boehringer Ingelheim Investigational Site, Jambes
  - 1237.6.32009 Boehringer Ingelheim Investigational Site, Lebbeke
  - 1237.6.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 1237.6.32006 Boehringer Ingelheim Investigational Site, Liège
  - 1237.6.32008 Boehringer Ingelheim Investigational Site, Ostend
  - 1237.6.32010 Boehringer Ingelheim Investigational Site, Turnhout
- Brazil (11):
  - 1237.6.55013 Boehringer Ingelheim Investigational Site, Botucatu
  - 1237.6.55010 Boehringer Ingelheim Investigational Site, Florianópolis
  - 1237.6.55012 Boehringer Ingelheim Investigational Site, Passo Fundo
  - 1237.6.55001 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.6.55002 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.6.55003 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.6.55005 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.6.55009 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1237.6.55006 Boehringer Ingelheim Investigational Site, São Paulo
  - 1237.6.55007 Boehringer Ingelheim Investigational Site, São Paulo
  - 1237.6.55011 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (11):
  - 1237.6.02109 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1237.6.02111 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1237.6.02106 Boehringer Ingelheim Investigational Site, Moncton, New Brunswick
  - 1237.6.02110 Boehringer Ingelheim Investigational Site, Courtice, Ontario
  - 1237.6.02101 Boehringer Ingelheim Investigational Site, Downsview, Ontario
  - 1237.6.02112 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1237.6.02103 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.6.02102 Boehringer Ingelheim Investigational Site, Windsor, Ontario
  - 1237.6.02104 Boehringer Ingelheim Investigational Site, Point Claire, Quebec
  - 1237.6.02105 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 1237.6.02108 Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
- China (16):
  - 1237.6.86117 Boehringer Ingelheim Investigational Site, Baotou
  - 1237.6.86102 Boehringer Ingelheim Investigational Site, Beijing
  - 1237.6.86104 Boehringer Ingelheim Investigational Site, Beijing
  - 1237.6.86105 Boehringer Ingelheim Investigational Site, Beijing
  - 1237.6.86115 Boehringer Ingelheim Investigational Site, Changsha
  - 1237.6.86110 Boehringer Ingelheim Investigational Site, Chengdu
  - 1237.6.86111 Boehringer Ingelheim Investigational Site, Chongqing
  - 1237.6.86109 Boehringer Ingelheim Investigational Site, Haikou
  - 1237.6.86108 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1237.6.86116 Boehringer Ingelheim Investigational Site, Hohhot
  - 1237.6.86114 Boehringer Ingelheim Investigational Site, Jinan
  - 1237.6.86106 Boehringer Ingelheim Investigational Site, Nanjing
  - 1237.6.86101 Boehringer Ingelheim Investigational Site, Shanghai
  - 1237.6.86113 Boehringer Ingelheim Investigational Site, Shenyang
  - 1237.6.86107 Boehringer Ingelheim Investigational Site, Suzhou
  - 1237.6.86112 Boehringer Ingelheim Investigational Site, Xi'an
- Colombia (6):
  - 1237.6.57001 Boehringer Ingelheim Investigational Site, Bogota DC
  - 1237.6.57003 Boehringer Ingelheim Investigational Site, Bogota DC
  - 1237.6.57007 Boehringer Ingelheim Investigational Site, Bogota DC
  - 1237.6.57008 Boehringer Ingelheim Investigational Site, Bogotá
  - 1237.6.57006 Boehringer Ingelheim Investigational Site, Cali
  - 1237.6.57004 Boehringer Ingelheim Investigational Site, Floridablanca
- Croatia (4):
  - 1237.6.38503 Boehringer Ingelheim Investigational Site, Petrinja
  - 1237.6.38504 Boehringer Ingelheim Investigational Site, Rijeka
  - 1237.6.38502 Boehringer Ingelheim Investigational Site, Zadar
  - 1237.6.38501 Boehringer Ingelheim Investigational Site, Zagreb
- Germany (13):
  - 1237.6.49022 Boehringer Ingelheim Investigational Site, Aschaffenburg
  - 1237.6.49017 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.6.49026 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.6.49027 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1237.6.49025 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1237.6.49016 Boehringer Ingelheim Investigational Site, Halle
  - 1237.6.49024 Boehringer Ingelheim Investigational Site, Hamburg
  - 1237.6.49021 Boehringer Ingelheim Investigational Site, Hanover
  - 1237.6.49019 Boehringer Ingelheim Investigational Site, Leipzig
  - 1237.6.49028 Boehringer Ingelheim Investigational Site, Mainz
  - 1237.6.49018 Boehringer Ingelheim Investigational Site, Rodgau/Dudenhofen
  - 1237.6.49020 Boehringer Ingelheim Investigational Site, Schwerin
  - 1237.6.49023 Boehringer Ingelheim Investigational Site, Teuchern
- Hungary (5):
  - 1237.6.36001 Boehringer Ingelheim Investigational Site, Debrecen
  - 1237.6.36004 Boehringer Ingelheim Investigational Site, Gödöllö
  - 1237.6.36005 Boehringer Ingelheim Investigational Site, Pécs
  - 1237.6.36003 Boehringer Ingelheim Investigational Site, Sopron
  - 1237.6.36002 Boehringer Ingelheim Investigational Site, Szeged
- India (8):
  - 1237.6.91003 Boehringer Ingelheim Investigational Site, Chennai
  - 1237.6.91011 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1237.6.91004 Boehringer Ingelheim Investigational Site, Jaipur
  - 1237.6.91002 Boehringer Ingelheim Investigational Site, Kolkata
  - 1237.6.91007 Boehringer Ingelheim Investigational Site, Maharastra
  - 1237.6.91006 Boehringer Ingelheim Investigational Site, Mumbai
  - 1237.6.91009 Boehringer Ingelheim Investigational Site, Nashik, Maharashtra
  - 1237.6.91008 Boehringer Ingelheim Investigational Site, Pune
- Ireland (3):
  - 1237.6.35304 Boehringer Ingelheim Investigational Site, County Limerick
  - 1237.6.35301 Boehringer Ingelheim Investigational Site, Dublin
  - 1237.6.35303 Boehringer Ingelheim Investigational Site, Dublin
- Japan (43):
  - 1237.6.81127 Boehringer Ingelheim Investigational Site, Abeno-ku, Osaka, Osaka
  - 1237.6.81123 Boehringer Ingelheim Investigational Site, Aoi-ku, Shizuoka, Shizuoka
  - 1237.6.81132 Boehringer Ingelheim Investigational Site, Chuo-ku, Kobe, Hyogo
  - 1237.6.81121 Boehringer Ingelheim Investigational Site, Fukui, Fukui
  - 1237.6.81137 Boehringer Ingelheim Investigational Site, Fukuyama, Hiroshima
  - 1237.6.81109 Boehringer Ingelheim Investigational Site, Hachioji, Tokyo
  - 1237.6.81134 Boehringer Ingelheim Investigational Site, Himeji, Hyogo
  - 1237.6.81106 Boehringer Ingelheim Investigational Site, Hitachi, Ibaraki
  - 1237.6.81139 Boehringer Ingelheim Investigational Site, Iizuka, Fukuoka
  - 1237.6.81102 Boehringer Ingelheim Investigational Site, Iwamizawa, Hokkaido
  - 1237.6.81117 Boehringer Ingelheim Investigational Site, Kamakura, Kanagawa
  - 1237.6.81120 Boehringer Ingelheim Investigational Site, Kanazawa, Ishikawa
  - 1237.6.81113 Boehringer Ingelheim Investigational Site, Kanazawa, Yokohama, Kanagawa
  - 1237.6.81108 Boehringer Ingelheim Investigational Site, Kashiwa, Chiba
  - 1237.6.81114 Boehringer Ingelheim Investigational Site, Kawasaki-ku, Kawasaki, Kanagawa
  - 1237.6.81135 Boehringer Ingelheim Investigational Site, Kita-ku, Okayama, Okayama
  - 1237.6.81126 Boehringer Ingelheim Investigational Site, Kita-ku, Sakai, Osaka
  - 1237.6.81101 Boehringer Ingelheim Investigational Site, Kita-ku, Sapporo, Hokkaido
  - 1237.6.81136 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 1237.6.81116 Boehringer Ingelheim Investigational Site, Minami-ku, Yokohama, Kanagawa
  - 1237.6.81118 Boehringer Ingelheim Investigational Site, Minami-ku, Yokohama, Kanagawa
  - 1237.6.81112 Boehringer Ingelheim Investigational Site, Mitaka, Tokyo
  - 1237.6.81105 Boehringer Ingelheim Investigational Site, Mito, Ibaraki
  - 1237.6.81142 Boehringer Ingelheim Investigational Site, Naha, Okinawa
  - 1237.6.81131 Boehringer Ingelheim Investigational Site, Nishi-ku, Kobe, Hyogo
  - 1237.6.81104 Boehringer Ingelheim Investigational Site, Obihiro, Hokkaido
  - 1237.6.81141 Boehringer Ingelheim Investigational Site, Okinawa, Okinawa
  - 1237.6.81110 Boehringer Ingelheim Investigational Site, Ota-ku, Tokyo
  - 1237.6.81138 Boehringer Ingelheim Investigational Site, Sakaide, Kagawa
  - 1237.6.81103 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1237.6.81140 Boehringer Ingelheim Investigational Site, Shimajiri-gun, Okinawa
  - 1237.6.81144 Boehringer Ingelheim Investigational Site, Shimajiri-gun, Okinawa
  - 1237.6.81111 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1237.6.81145 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1237.6.81107 Boehringer Ingelheim Investigational Site, Soka, Saitama
  - 1237.6.81133 Boehringer Ingelheim Investigational Site, Takarazuka, Hyogo
  - 1237.6.81122 Boehringer Ingelheim Investigational Site, Takayama, Gifu
  - 1237.6.81143 Boehringer Ingelheim Investigational Site, Tomigusuku, Okinawa
  - 1237.6.81128 Boehringer Ingelheim Investigational Site, Toyonaka, Osaka
  - 1237.6.81124 Boehringer Ingelheim Investigational Site, Uji, Kyoto
  - 1237.6.81130 Boehringer Ingelheim Investigational Site, Yabu, Hyogo
  - 1237.6.81129 Boehringer Ingelheim Investigational Site, Yao, Osaka
  - 1237.6.81119 Boehringer Ingelheim Investigational Site, Yokosuka, Kanagawa
- Norway (7):
  - 1237.6.47005 Boehringer Ingelheim Investigational Site, Elverum
  - 1237.6.47001 Boehringer Ingelheim Investigational Site, Hønefoss
  - 1237.6.47002 Boehringer Ingelheim Investigational Site, Kløfta
  - 1237.6.47004 Boehringer Ingelheim Investigational Site, Lierskogen
  - 1237.6.47003 Boehringer Ingelheim Investigational Site, Oslo
  - 1237.6.47007 Boehringer Ingelheim Investigational Site, Ski
  - 1237.6.47008 Boehringer Ingelheim Investigational Site, Svelvik
- Romania (5):
  - 1237.6.40004 Boehringer Ingelheim Investigational Site, Arad
  - 1237.6.40005 Boehringer Ingelheim Investigational Site, Arad
  - 1237.6.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1237.6.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1237.6.40003 Boehringer Ingelheim Investigational Site, Cluj-Napoca
- Russia (5):
  - 1237.6.07004 Boehringer Ingelheim Investigational Site, Moscow
  - 1237.6.07005 Boehringer Ingelheim Investigational Site, Moscow
  - 1237.6.07002 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.6.07003 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1237.6.07001 Boehringer Ingelheim Investigational Site, Yaroslavl
- Serbia (5):
  - 1237.6.38103 Boehringer Ingelheim Investigational Site, Belgrade
  - 1237.6.38104 Boehringer Ingelheim Investigational Site, Belgrade
  - 1237.6.38105 Boehringer Ingelheim Investigational Site, Belgrade
  - 1237.6.38102 Boehringer Ingelheim Investigational Site, Kragujevac
  - 1237.6.38101 Boehringer Ingelheim Investigational Site, Niš
- Slovakia (6):
  - 1237.6.42101 Boehringer Ingelheim Investigational Site, Bardejov
  - 1237.6.42102 Boehringer Ingelheim Investigational Site, Bojnice
  - 1237.6.42104 Boehringer Ingelheim Investigational Site, Košice
  - 1237.6.42107 Boehringer Ingelheim Investigational Site, Nitra
  - 1237.6.42103 Boehringer Ingelheim Investigational Site, Spišská Nová Ves
  - 1237.6.42106 Boehringer Ingelheim Investigational Site, Žilina
- South Africa (5):
  - 1237.6.27002 Boehringer Ingelheim Investigational Site, Bellville
  - 1237.6.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.6.27003 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.6.27004 Boehringer Ingelheim Investigational Site, Cape Town
  - 1237.6.27005 Boehringer Ingelheim Investigational Site, Pretoria
- Spain (8):
  - 1237.6.34008 Boehringer Ingelheim Investigational Site, Badalona (Barcelona)
  - 1237.6.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 1237.6.34009 Boehringer Ingelheim Investigational Site, Barcelona
  - 1237.6.34001 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 1237.6.34002 Boehringer Ingelheim Investigational Site, Mérida
  - 1237.6.34005 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
  - 1237.6.34004 Boehringer Ingelheim Investigational Site, Sant Joan d'Alacant
  - 1237.6.34006 Boehringer Ingelheim Investigational Site, Vic (Barcelona)
- Sweden (7):
  - 1237.6.46003 Boehringer Ingelheim Investigational Site, Boden
  - 1237.6.46002 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1237.6.46006 Boehringer Ingelheim Investigational Site, Härnösand
  - 1237.6.46005 Boehringer Ingelheim Investigational Site, Höllviken
  - 1237.6.46001 Boehringer Ingelheim Investigational Site, Lund
  - 1237.6.46004 Boehringer Ingelheim Investigational Site, Stockholm
  - 1237.6.46007 Boehringer Ingelheim Investigational Site, Uddevalla
- Taiwan (7):
  - 1237.6.88607 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1237.6.88608 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1237.6.88602 Boehringer Ingelheim Investigational Site, New Taipei City
  - 1237.6.88604 Boehringer Ingelheim Investigational Site, Taichung
  - 1237.6.88605 Boehringer Ingelheim Investigational Site, Tainan
  - 1237.6.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 1237.6.88603 Boehringer Ingelheim Investigational Site, Taoyuan
- Turkey (Türkiye) (5):
  - 1237.6.90105 Boehringer Ingelheim Investigational Site, Ankara
  - 1237.6.90103 Boehringer Ingelheim Investigational Site, Denizli
  - 1237.6.90104 Boehringer Ingelheim Investigational Site, Istanbul
  - 1237.6.90101 Boehringer Ingelheim Investigational Site, Izmir
  - 1237.6.90102 Boehringer Ingelheim Investigational Site, Izmir
- United Kingdom (7):
  - 1237.6.44002 Boehringer Ingelheim Investigational Site, Blackpool
  - 1237.6.44009 Boehringer Ingelheim Investigational Site, Blackpool
  - 1237.6.44007 Boehringer Ingelheim Investigational Site, Bristol
  - 1237.6.44010 Boehringer Ingelheim Investigational Site, Chertsey
  - 1237.6.44011 Boehringer Ingelheim Investigational Site, Fleetwood
  - 1237.6.44001 Boehringer Ingelheim Investigational Site, Manchester
  - 1237.6.44008 Boehringer Ingelheim Investigational Site, Midsomer Norton

REFERENCES:
- [Derived] Rabe KF, Chalmers JD, Miravitlles M, Kocks JWH, Tsiligianni I, de la Hoz A, Xue W, Singh D, Ferguson GT, Wedzicha J. Tiotropium/Olodaterol Delays Clinically Important Deterioration Compared with Tiotropium Monotherapy in Patients with Early COPD: a Post Hoc Analysis of the TONADO(R) Trials. Adv Ther. 2021 Jan;38(1):579-593. doi: 10.1007/s12325-020-01528-2. Epub 2020 Nov 11. PMID 33175291
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Andreas S, Bothner U, de la Hoz A, Kloer I, Trampisch M, Alter P. No Influence on Cardiac Arrhythmia or Heart Rate from Long-Term Treatment with Tiotropium/Olodaterol versus Monocomponents by Holter ECG Analysis in Patients with Moderate-to-Very-Severe COPD. Int J Chron Obstruct Pulmon Dis. 2020 Aug 10;15:1945-1953. doi: 10.2147/COPD.S246350. eCollection 2020. PMID 32848380
- [Derived] Andreas S, McGarvey L, Bothner U, Trampisch M, de la Hoz A, Flezar M, Buhl R, Alter P. Absence of Adverse Effects of Tiotropium/Olodaterol Compared with the Monocomponents on Long-Term Heart Rate and Blood Pressure in Patients with Moderate-to-Very-Severe COPD. Int J Chron Obstruct Pulmon Dis. 2020 Aug 10;15:1935-1944. doi: 10.2147/COPD.S246348. eCollection 2020. PMID 32848379
- [Derived] Wedzicha JA, Buhl R, Singh D, Vogelmeier CF, de la Hoz A, Xue W, Anzueto A, Calverley PMA. Tiotropium/Olodaterol Decreases Exacerbation Rates Compared with Tiotropium in a Range of Patients with COPD: Pooled Analysis of the TONADO(R)/DYNAGITO(R) Trials. Adv Ther. 2020 Oct;37(10):4266-4279. doi: 10.1007/s12325-020-01438-3. Epub 2020 Aug 10. PMID 32776202
- [Derived] Buhl R, de la Hoz A, Xue W, Singh D, Ferguson GT. Efficacy of Tiotropium/Olodaterol Compared with Tiotropium as a First-Line Maintenance Treatment in Patients with COPD Who Are Naive to LAMA, LABA and ICS: Pooled Analysis of Four Clinical Trials. Adv Ther. 2020 Oct;37(10):4175-4189. doi: 10.1007/s12325-020-01411-0. Epub 2020 Jul 15. PMID 32671684
- [Derived] Buhl R, Singh D, de la Hoz A, Xue W, Ferguson GT. Benefits of Tiotropium/Olodaterol Compared with Tiotropium in Patients with COPD Receiving only LAMA at Baseline: Pooled Analysis of the TONADO(R) and OTEMTO(R) Studies. Adv Ther. 2020 Aug;37(8):3485-3499. doi: 10.1007/s12325-020-01373-3. Epub 2020 May 27. PMID 32462607
- [Derived] Ferguson GT, Buhl R, Bothner U, Hoz A, Voss F, Anzueto A, Calverley PMA. Safety of tiotropium/olodaterol in chronic obstructive pulmonary disease: pooled analysis of three large, 52-week, randomized clinical trials. Respir Med. 2018 Oct;143:67-73. doi: 10.1016/j.rmed.2018.08.012. Epub 2018 Aug 28. PMID 30261995
- [Derived] Maltais F, Buhl R, Koch A, Amatto VC, Reid J, Gronke L, Bothner U, Voss F, McGarvey L, Ferguson GT. beta-Blockers in COPD: A Cohort Study From the TONADO Research Program. Chest. 2018 Jun;153(6):1315-1325. doi: 10.1016/j.chest.2018.01.008. Epub 2018 Jan 31. PMID 29355547
- [Derived] Buhl R, Magder S, Bothner U, Tetzlaff K, Voss F, Loaiza L, Vogelmeier CF, McGarvey L. Long-term general and cardiovascular safety of tiotropium/olodaterol in patients with moderate to very severe chronic obstructive pulmonary disease. Respir Med. 2017 Jan;122:58-66. doi: 10.1016/j.rmed.2016.11.011. Epub 2016 Nov 14. PMID 27993292
- [Derived] Ferguson GT, Flezar M, Korn S, Korducki L, Gronke L, Abrahams R, Buhl R. Efficacy of Tiotropium + Olodaterol in Patients with Chronic Obstructive Pulmonary Disease by Initial Disease Severity and Treatment Intensity: A Post Hoc Analysis. Adv Ther. 2015 Jun;32(6):523-36. doi: 10.1007/s12325-015-0218-0. Epub 2015 Jun 26. PMID 26112656
- [Derived] Buhl R, Maltais F, Abrahams R, Bjermer L, Derom E, Ferguson G, Flezar M, Hebert J, McGarvey L, Pizzichini E, Reid J, Veale A, Gronke L, Hamilton A, Korducki L, Tetzlaff K, Waitere-Wijker S, Watz H, Bateman E. Tiotropium and olodaterol fixed-dose combination versus mono-components in COPD (GOLD 2-4). Eur Respir J. 2015 Apr;45(4):969-79. doi: 10.1183/09031936.00136014. Epub 2015 Jan 8. PMID 25573406

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial was one of 2 confirmatory Phase III 52-week, multi-centre, multi-national, randomised, double-blind, parallel group studies to evaluate the long-term efficacy and safety of once daily treatment with orally inhaled Tio+Olo FDC (2.5/5μg; 5/5μg) compared with the individual components (2.5μg; 5μg Tiotropium, 5μg Olodaterol) in COPD patients
Groups:
- Olodaterol (5 μg): Oral inhalation of Olodaterol 5 μg (2.5 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tiotropium (2.5 μg): Oral inhalation of Tiotropium 2.5 μg (1.25 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tiotropium (5 μg): Oral inhalation of Tiotropium 5 μg (2.5 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tio+Olo FDC (2.5/5 μg): Oral inhalation of fixed dose combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg (Tiotropium: 1.25 μg per actuation and Olodaterol: 2.5 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tio+Olo FDC (5/5 μg): Oral inhalation of FDC of Tiotropium 5 μg and Olodaterol 5 μg (Tiotropium and Olodaterol: 2.5 μg per actuation), 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
Period: Overall Study
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Started | 510 (started are actually the randomized) | 507 | 507 | 508 | 507
Completed | 412 | 409 | 410 | 445 | 430
Not Completed | 98 | 98 | 97 | 63 | 77
Not completed — not treated | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 59 | 57 | 53 | 33 | 41
Not completed — Non compliant with protocol | 6 | 6 | 5 | 6 | 5
Not completed — Lost to Follow-up | 0 | 3 | 2 | 3 | 1
Not completed — Consent withdrawn not due to AE | 29 | 30 | 34 | 19 | 29
Not completed — not stated above | 4 | 2 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all patients in the randomised set who were dispensed study medication and were documented to have taken any dose of study medication.
Groups:
- Olodaterol (5 μg): Oral inhalation of Olodaterol 5 μg (2.5 μg per actuation), 2 puffs in the morning.
- Tiotropium (2.5 μg): Oral inhalation of Tiotropium 2.5 μg (1.25 μg per actuation), 2 puffs in the morning.
- Tiotropium (5 μg): Oral inhalation of Tiotropium 5 μg (2.5 μg per actuation), 2 puffs in the morning.
- Tio+Olo FDC (2.5/5 μg): Oral inhalation of FDC of Tiotropium 2.5 μg and Olodaterol 5 μg (Tiotropium: 1.25 μg per actuation and Olodaterol: 2.5 μg per actuation), 2 puffs in the morning.
- Tio+Olo FDC (5/5 μg): Oral inhalation of FDC of Tiotropium 5 μg and Olodaterol 5 μg (Tiotropium and Olodaterol: 2.5 μg per actuation), 2 puffs in the morning.
- Total: Total of all reporting groups
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg) | Total
Number analyzed (Participants) | 510 | 507 | 506 | 508 | 507 | 2538
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (8.3) | 63.9 (8.7) | 63.5 (8.7) | 64.1 (7.6) | 62.7 (8.4) | 63.8 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 146 | 134 | 140 | 158 | 710
  Male | 378 | 361 | 372 | 368 | 349 | 1828

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) (0-3h) Response on Day 169
Description: FEV1 AUC(0-3h) was calculated as the area under the FEV1- time curve from 0 to 3 h post-dose using the trapezoidal rule, divided by the duration (3 h) to report in litres. FEV1 AUC(0-3h) response was defined as FEV1 AUC(0-3h) minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom. Number of participants analyzed are the number of patients contributing to the MMRM model in each treatment group.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 169 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h post-dose on Day 169
Population: The Full analysis set (FAS) included all patients who were randomised, who were dispensed study medication, were documented to have taken any dose of study medication and who had a non-missing baseline and at least one non-missing post-baseline measurement before or at Week 24 for any of the primary and key secondary efficacy endpoints.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 507 | 504 | 500 | 506 | 502
Litres | 0.136 (0.009) | 0.125 (0.009) | 0.165 (0.009) | 0.256 (0.009) | 0.268 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.132, 95% CI 2-sided [0.108 to 0.157], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.103, 95% CI 2-sided [0.078 to 0.127], Standard Error of Mean 0.012 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.121, 95% CI 2-sided [0.096 to 0.145], Standard Error of Mean 0.012 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.131, 95% CI 2-sided [0.106 to 0.155], Standard Error of Mean 0.012 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.091, 95% CI 2-sided [0.066 to 0.115], Standard Error of Mean 0.012 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.3394, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.012, 95% CI 2-sided [-0.013 to 0.036], Standard Error of Mean 0.012 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.143, 95% CI 2-sided [0.118 to 0.167], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0173, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.030, 95% CI 2-sided [0.005 to 0.054], Standard Error of Mean 0.012 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.4210, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.010, 95% CI 2-sided [-0.035 to 0.014], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.040, 95% CI 2-sided [0.015 to 0.064], Standard Error of Mean 0.012 — spatial power covariance structure for within-patient errors

2. Primary Outcome: Trough FEV1 Response on Day 170
Description: Trough FEV1 was defined as the FEV1 value at the end of the dosing interval (24 hours) and was calculated as the mean of the 2 FEV1 measurements performed at 23 h and at 23 h 50 min after inhalation of study medication at the clinic visit on the previous day.
  Trough FEV1 response was defined as trough FEV1 minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an MMRM including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 23 h and at 23 h 50 min after inhalation of study medication on Day 170
Population: FAS. Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.057 (0.009) | 0.062 (0.009) | 0.096 (0.009) | 0.125 (0.009) | 0.145 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.088, 95% CI 2-sided [0.063 to 0.113], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.050, 95% CI 2-sided [0.024 to 0.075], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.067, 95% CI 2-sided [0.042 to 0.092], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.062, 95% CI 2-sided [0.037 to 0.087], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0231, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.029, 95% CI 2-sided [0.004 to 0.054], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1073, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.021, 95% CI 2-sided [-0.004 to 0.046], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.083, 95% CI 2-sided [0.058 to 0.108], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0029, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.038, 95% CI 2-sided [0.013 to 0.063], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.6939, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.005, 95% CI 2-sided [-0.020 to 0.030], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0097, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.033, 95% CI 2-sided [0.008 to 0.058], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors

3. Primary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score on Day 169 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274).
Description: The SGRQ is designed to measure health impairment in patients with COPD. It is divided into 2 parts: part 1 produces the symptoms score, and part 2 the activity and impacts scores. A total score is also produced. Each subscale score is the sum of the weights for the items in the subscale as a percent of the sum of the weights for a patient in the worst possible condition. The total score uses the same calculation except that the weights are summed over the entire questionnaire. The individual subscales as well as the total score can range from 0 to 100 with a lower score denoting a better health status.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 169
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 954 | 960 | 954 | 990 | 979
points on a scale | 38.366 (0.396) | 37.792 (0.390) | 37.907 (0.393) | 37.335 (0.385) | 36.674 (0.386)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.693, 95% CI 2-sided [-2.778 to -0.608], Standard Error of Mean 0.553 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0252, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.233, 95% CI 2-sided [-2.313 to -0.153], Standard Error of Mean 0.551 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0620, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.031, 95% CI 2-sided [-2.113 to 0.052], Standard Error of Mean 0.552 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.4051, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.456, 95% CI 2-sided [-1.531 to 0.618], Standard Error of Mean 0.548 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.2988, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.571, 95% CI 2-sided [-1.649 to 0.507], Standard Error of Mean 0.550 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2249, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.662, 95% CI 2-sided [-1.731 to 0.407], Standard Error of Mean 0.545 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0418, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.118, 95% CI 2-sided [-2.195 to -0.042], Standard Error of Mean 0.549 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4097, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.460, 95% CI 2-sided [-1.552 to 0.633], Standard Error of Mean 0.557 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.3013, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.575, 95% CI 2-sided [-1.664 to 0.515], Standard Error of Mean 0.556 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8355, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.115, 95% CI 2-sided [-0.970 to 1.200], Standard Error of Mean 0.554 — spatial power covariance structure for within-patient errors

4. Secondary Outcome: Mahler Transitional Dyspnoea Index (TDI) Focal Score on Day 169 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: Mahler Transitional Dyspnoea Index (TDI) focal score on Day 169 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274) is the key secondary endpoint.
  The Mahler Dyspnoea questionnaire is an instrument which measures change from the baseline state The TDI focal score was used to measure the effect of Tio+Olo FDC on patients' dyspnoea after 24 weeks of treatment (Day 169). The focal score is the sum of the subscale scores for Functional Impairment, Magnitude of Effort and Magnitude of Task. Scores for each subscale range from -3 to 3 so that the Focal score ranges from -9 to 9. For all subscale scores and the Focal score a higher value indicates a better outcome.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 169
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 984 | 982 | 978 | 992 | 992
points on a scale | 1.564 (0.096) | 1.690 (0.095) | 1.627 (0.096) | 1.980 (0.095) | 1.983 (0.095)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.420, 95% CI 2-sided [0.155 to 0.684], Standard Error of Mean 0.135 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0082, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.356, 95% CI 2-sided [0.092 to 0.619], Standard Error of Mean 0.135 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.416, 95% CI 2-sided [0.152 to 0.681], Standard Error of Mean 0.135 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0307, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.290, 95% CI 2-sided [0.027 to 0.554], Standard Error of Mean 0.134 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0088, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.352, 95% CI 2-sided [0.089 to 0.616], Standard Error of Mean 0.135 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.9801, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.003, 95% CI 2-sided [-0.259 to 0.266], Standard Error of Mean 0.134 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0289, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.294, 95% CI 2-sided [0.030 to 0.557], Standard Error of Mean 0.134 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6382, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.064, 95% CI 2-sided [-0.202 to 0.330], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.3525, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.126, 95% CI 2-sided [-0.140 to 0.391], Standard Error of Mean 0.135 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6457, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.062, 95% CI 2-sided [-0.327 to 0.203], Standard Error of Mean 0.135 — Spatial power covariance structure for within-patient errors

5. Secondary Outcome: FEV1 AUC(0-3h) Response on Day 1
Description: FEV1 AUC(0-3h) was calculated as the area under the FEV1- time curve from 0 to 3 h post-dose using the trapezoidal rule, divided by the duration (3 h) to report in litres.
  FEV1 AUC(0-3h) response was defined as FEV1 AUC(0-3h) minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose of randomised treatment at Day1.
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to 5 min, 15 min, 30 min, 1 h, 2 h, 3 h post-dose on the first day of randomized treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 507 | 504 | 500 | 506 | 502
Litres | 0.196 (0.009) | 0.135 (0.009) | 0.164 (0.009) | 0.228 (0.009) | 0.229 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0095, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.033, 95% CI 2-sided [0.008 to 0.058], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.065, 95% CI 2-sided [0.040 to 0.090], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0112, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.033, 95% CI 2-sided [0.007 to 0.058], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.093, 95% CI 2-sided [0.068 to 0.119], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.064, 95% CI 2-sided [0.039 to 0.090], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.9514, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.001, 95% CI 2-sided [-0.024 to 0.026], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.094, 95% CI 2-sided [0.069 to 0.119], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0131, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.032, 95% CI 2-sided [-0.057 to -0.007], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.061, 95% CI 2-sided [-0.086 to -0.036], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0243, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.029, 95% CI 2-sided [0.004 to 0.054], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors

6. Secondary Outcome: FEV1 AUC(0-3h) Response on Day 85
Description: as for outcome 5
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 85 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h post-dose on Day 85
Population: FAS (on day 85). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 507 | 504 | 500 | 506 | 502
Litres | 0.153 (0.009) | 0.165 (0.009) | 0.187 (0.009) | 0.272 (0.009) | 0.297 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.145, 95% CI 2-sided [0.119 to 0.170], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.111, 95% CI 2-sided [0.085 to 0.136], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.119, 95% CI 2-sided [0.094 to 0.144], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.106, 95% CI 2-sided [0.081 to 0.132], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.085, 95% CI 2-sided [0.059 to 0.110], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0470, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.026, 95% CI 2-sided [0.000 to 0.051], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.132, 95% CI 2-sided [0.107 to 0.158], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0083, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.034, 95% CI 2-sided [0.009 to 0.060], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.3329, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.013, 95% CI 2-sided [-0.013 to 0.038], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0958, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.022, 95% CI 2-sided [-0.004 to 0.047], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors

7. Secondary Outcome: FEV1 AUC(0-3h) Response on Day 365
Description: as for outcome 5
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 365 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h post-dose on Day 365
Population: FAS (on day 365). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 507 | 504 | 500 | 506 | 502
Litres | 0.105 (0.010) | 0.105 (0.010) | 0.124 (0.010) | 0.223 (0.009) | 0.237 (0.010)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.132, 95% CI 2-sided [0.105 to 0.158], Standard Error of Mean 0.014 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.112, 95% CI 2-sided [0.086 to 0.139], Standard Error of Mean 0.014 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.118, 95% CI 2-sided [0.092 to 0.144], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.118, 95% CI 2-sided [0.092 to 0.144], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.098, 95% CI 2-sided [0.072 to 0.125], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.3008, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.014, 95% CI 2-sided [-0.012 to 0.040], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.132, 95% CI 2-sided [0.105 to 0.158], Standard Error of Mean 0.014 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1484, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.020, 95% CI 2-sided [-0.007 to 0.046], Standard Error of Mean 0.014 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.9981, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.000, 95% CI 2-sided [-0.026 to 0.027], Standard Error of Mean 0.014 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1480, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.020, 95% CI 2-sided [-0.007 to 0.046], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors

8. Secondary Outcome: Trough FEV1 Response on Day 15
Description: Trough FEV1 was defined as the FEV1 value at the end of the dosing interval (24 hours), calculated as the mean of the pre-dose measurements.
  Trough FEV1 response was defined as trough FEV1 minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose of randomised treatment at Day1.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 10 min pre-dose on day 15
Population: FAS (day 15). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.083 (0.009) | 0.085 (0.009) | 0.112 (0.009) | 0.147 (0.009) | 0.148 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.065, 95% CI 2-sided [0.040 to 0.090], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0050, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.036, 95% CI 2-sided [0.011 to 0.061], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.064, 95% CI 2-sided [0.039 to 0.089], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.063, 95% CI 2-sided [0.037 to 0.088], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0057, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.036, 95% CI 2-sided [0.010 to 0.061], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.9633, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.001, 95% CI 2-sided [-0.025 to 0.026], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.063, 95% CI 2-sided [0.038 to 0.088], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0250, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.029, 95% CI 2-sided [0.004 to 0.054], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.8949, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.002, 95% CI 2-sided [-0.023 to 0.027], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0351, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.027, 95% CI 2-sided [0.002 to 0.052], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors

9. Secondary Outcome: Trough FEV1 Response on Day 43
Description: as for outcome 8
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 10 min pre-dose on day 43
Population: FAS (day 43). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.070 (0.009) | 0.085 (0.009) | 0.103 (0.009) | 0.146 (0.009) | 0.150 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.080, 95% CI 2-sided [0.055 to 0.105], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.047, 95% CI 2-sided [0.022 to 0.073], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.076, 95% CI 2-sided [0.051 to 0.101], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.061, 95% CI 2-sided [0.036 to 0.086], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.044, 95% CI 2-sided [0.018 to 0.069], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.7755, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.004, 95% CI 2-sided [-0.022 to 0.029], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.065, 95% CI 2-sided [0.039 to 0.090], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0118, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.032, 95% CI 2-sided [0.007 to 0.058], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.2416, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.015, 95% CI 2-sided [-0.010 to 0.040], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1792, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.017, 95% CI 2-sided [-0.008 to 0.043], Standard Error of Mean 0.013 — Spatial power covariance structure for within-patient errors

10. Secondary Outcome: Trough FEV1 Response on Day 85
Description: as for outcome 8
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 1hr and 10 min pre-dose on day 85
Population: FAS (day 85). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.047 (0.009) | 0.081 (0.009) | 0.088 (0.009) | 0.129 (0.009) | 0.147 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.100, 95% CI 2-sided [0.074 to 0.125], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.059, 95% CI 2-sided [0.033 to 0.084], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.082, 95% CI 2-sided [0.057 to 0.107], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.048, 95% CI 2-sided [0.023 to 0.073], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.041, 95% CI 2-sided [0.016 to 0.067], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1747, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.018, 95% CI 2-sided [-0.008 to 0.043], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.065, 95% CI 2-sided [0.040 to 0.091], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0016, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.041, 95% CI 2-sided [0.016 to 0.066], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0081, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.034, 95% CI 2-sided [0.009 to 0.060], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6110, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.007, 95% CI 2-sided [-0.019 to 0.032], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors

11. Secondary Outcome: Trough FEV1 Response on Day 169
Description: as for outcome 8
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 1hr and 10 min pre-dose on day 169
Population: FAS (day 169). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.034 (0.009) | 0.041 (0.009) | 0.068 (0.009) | 0.111 (0.009) | 0.119 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.085, 95% CI 2-sided [0.059 to 0.111], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.050, 95% CI 2-sided [0.025 to 0.076], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.077, 95% CI 2-sided [0.051 to 0.102], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.069, 95% CI 2-sided [0.044 to 0.095], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.042, 95% CI 2-sided [0.016 to 0.068], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.5274, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.008, 95% CI 2-sided [-0.017 to 0.034], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.078, 95% CI 2-sided [0.052 to 0.103], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0083, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.035, 95% CI 2-sided [0.009 to 0.060], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.5744, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.007, 95% CI 2-sided [-0.018 to 0.033], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0381, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.027, 95% CI 2-sided [0.001 to 0.053], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors

12. Secondary Outcome: Trough FEV1 Response on Day 365
Description: as for outcome 8
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 1 hr and 10 min pre-dose on day 365
Population: FAS (day 365). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.011 (0.009) | 0.022 (0.009) | 0.040 (0.009) | 0.077 (0.009) | 0.093 (0.009)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.081, 95% CI 2-sided [0.055 to 0.108], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.053, 95% CI 2-sided [0.027 to 0.079], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.065, 95% CI 2-sided [0.039 to 0.091], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.055, 95% CI 2-sided [0.029 to 0.081], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0052, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.037, 95% CI 2-sided [0.011 to 0.063], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2273, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.016, 95% CI 2-sided [-0.010 to 0.042], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.071, 95% CI 2-sided [0.045 to 0.097], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0330, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.028, 95% CI 2-sided [0.002 to 0.055], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.4327, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.010, 95% CI 2-sided [-0.016 to 0.037], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1764, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.018, 95% CI 2-sided [-0.008 to 0.044], Standard Error of Mean 0.013 — spatial power covariance structure for within-patient errors

13. Secondary Outcome: Forced Vital Capacity (FVC) AUC(0-3h) Response on Day 1
Description: FVC AUC(0-3h) was calculated as the area under the FVC- time curve from 0 to 3 h post-dose using the trapezoidal rule, divided by the duration (3 h) to report in litres.
  FVC AUC(0-3h) response was defined as FVC AUC(0-3h) minus baseline FVC.Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: as for outcome 5
Population: FAS (day 1). Since it is possible for the patient to meet the data criterion for only a subset of the primary endpoints, it is possible that the number of patients used in the FAS analysis for different endpoints will vary.
Measure: Median (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 507 | 504 | 500 | 506 | 502
Litres | 0.341 (0.018) | 0.264 (0.018) | 0.298 (0.018) | 0.411 (0.018) | 0.397 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0241, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.056, 95% CI 2-sided [0.007 to 0.105], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.100, 95% CI 2-sided [0.051 to 0.148], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0049, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.070, 95% CI 2-sided [0.021 to 0.119], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.147, 95% CI 2-sided [0.098 to 0.196], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.113, 95% CI 2-sided [0.064 to 0.162], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.5831, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.014, 95% CI 2-sided [-0.063 to 0.035], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.133, 95% CI 2-sided [0.084 to 0.182], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0822, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.043, 95% CI 2-sided [-0.092 to 0.006], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0020, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.077, 95% CI 2-sided [-0.126 to -0.028], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1774, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.034, 95% CI 2-sided [-0.015 to 0.083], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors

14. Secondary Outcome: Forced Vital Capacity (FVC) AUC(0-3h) Response on Day 85
Description: as for outcome 13
Time Frame: as for outcome 6
Population: as for outcome 10
Measure: Median (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 507 | 504 | 500 | 506 | 502
Litres | 0.250 (0.018) | 0.306 (0.018) | 0.326 (0.018) | 0.460 (0.018) | 0.469 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.219, 95% CI 2-sided [0.169 to 0.268], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.143, 95% CI 2-sided [0.094 to 0.193], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.209, 95% CI 2-sided [0.160 to 0.258], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.153, 95% CI 2-sided [0.104 to 0.203], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.134, 95% CI 2-sided [0.084 to 0.183], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.6974, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.010, 95% CI 2-sided [-0.040 to 0.059], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.163, 95% CI 2-sided [0.114 to 0.213], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0027, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.076, 95% CI 2-sided [0.026 to 0.125], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0269, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.056, 95% CI 2-sided [0.006 to 0.105], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4343, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.020, 95% CI 2-sided [-0.030 to 0.069], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors

15. Secondary Outcome: Forced Vital Capacity (FVC) AUC(0-3h) Response on Day 169
Description: FVC AUC(0-3h) was calculated as the area under the FVC- time curve from 0 to 3 h post-dose using the trapezoidal rule, divided by the duration (3 h) to report in litres.
  FVC AUC(0-3h) response was defined as FVC AUC(0-3h) minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Median (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 507 | 504 | 500 | 506 | 502
Litres | 0.231 (0.018) | 0.247 (0.018) | 0.283 (0.018) | 0.439 (0.018) | 0.429 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.198, 95% CI 2-sided [0.148 to 0.248], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.146, 95% CI 2-sided [0.096 to 0.197], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.208, 95% CI 2-sided [0.158 to 0.258], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.193, 95% CI 2-sided [0.143 to 0.242], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.156, 95% CI 2-sided [0.106 to 0.206], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.6980, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.010, 95% CI 2-sided [-0.060 to 0.040], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.183, 95% CI 2-sided [0.132 to 0.233], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0442, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.051, 95% CI 2-sided [0.001 to 0.102], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.5514, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.015, 95% CI 2-sided [-0.035 to 0.065], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1569, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.036, 95% CI 2-sided [-0.014 to 0.086], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors

16. Secondary Outcome: Forced Vital Capacity (FVC) AUC(0-3h) Response on Day 365
Description: as for outcome 15
Time Frame: as for outcome 7
Population: as for outcome 12
Measure: Median (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 507 | 504 | 500 | 506 | 502
Litres | 0.180 (0.019) | 0.216 (0.018) | 0.198 (0.019) | 0.397 (0.018) | 0.381 (0.019)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.202, 95% CI 2-sided [0.150 to 0.253], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.183, 95% CI 2-sided [0.132 to 0.234], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.218, 95% CI 2-sided [0.167 to 0.269], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day^interaction; patient as a random effect; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.181, 95% CI 2-sided [0.130 to 0.232], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.199, 95% CI 2-sided [0.148 to 0.250], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.5373, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.016, 95% CI 2-sided [-0.067 to 0.035], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.165, 95% CI 2-sided [0.114 to 0.216], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4763, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.019, 95% CI 2-sided [-0.033 to 0.070], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1613, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.037, 95% CI 2-sided [-0.015 to 0.088], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4908, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.018, 95% CI 2-sided [-0.069 to 0.033], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors

17. Secondary Outcome: Trough FVC Response on Day 15
Description: Trough FVC was defined as the FVC value at the end of the dosing interval (24 hours), calculated as the mean of the pre-dose measurements.
  Trough FVC response was defined as trough FVC minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
  The adjusted means (SE) were obtained from fitting an Mixed effect model repeated measures (MMRM) including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 10 min pre-dose on day 15
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.163 (0.018) | 0.209 (0.018) | 0.222 (0.018) | 0.293 (0.018) | 0.285 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.122, 95% CI 2-sided [0.072 to 0.173], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0154, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.063, 95% CI 2-sided [0.012 to 0.113], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.130, 95% CI 2-sided [0.080 to 0.181], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0012, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.084, 95% CI 2-sided [0.033 to 0.134], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0061, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.071, 95% CI 2-sided [0.020 to 0.121], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.7518, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.008, 95% CI 2-sided [-0.059 to 0.042], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0034, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.076, 95% CI 2-sided [0.025 to 0.126], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0209, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.059, 95% CI 2-sided [0.009 to 0.110], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0708, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.047, 95% CI 2-sided [-0.004 to 0.097], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6148, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.013, 95% CI 2-sided [-0.038 to 0.064], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors

18. Secondary Outcome: Trough FVC Response on Day 43
Description: as for outcome 17
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 10 min pre-dose on day 43
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.129 (0.018) | 0.206 (0.018) | 0.222 (0.018) | 0.281 (0.018) | 0.293 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.164, 95% CI 2-sided [0.114 to 0.215], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0064, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.071, 95% CI 2-sided [0.020 to 0.122], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.152, 95% CI 2-sided [0.102 to 0.203], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0035, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.075, 95% CI 2-sided [0.025 to 0.126], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0233, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.059, 95% CI 2-sided [0.008 to 0.109], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.6413, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.012, 95% CI 2-sided [-0.039 to 0.063], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.088, 95% CI 2-sided [0.037 to 0.138], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.094, 95% CI 2-sided [0.043 to 0.144], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0030, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.077, 95% CI 2-sided [0.026 to 0.127], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.5159, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.017, 95% CI 2-sided [-0.034 to 0.068], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors

19. Secondary Outcome: Trough FVC Response on Day 85
Description: as for outcome 17
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and on day 85
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.063 (0.018) | 0.178 (0.018) | 0.184 (0.018) | 0.246 (0.018) | 0.274 (0.019)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.210, 95% CI 2-sided [0.159 to 0.261], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.089, 95% CI 2-sided [0.038 to 0.141], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.183, 95% CI 2-sided [0.132 to 0.234], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0094, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.068, 95% CI 2-sided [0.017 to 0.119], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0174, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.062, 95% CI 2-sided [0.011 to 0.113], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2888, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.028, 95% CI 2-sided [-0.023 to 0.079], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0003, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.095, 95% CI 2-sided [0.044 to 0.146], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.121, 95% CI 2-sided [0.070 to 0.172], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.115, 95% CI 2-sided [0.064 to 0.166], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8241, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.006, 95% CI 2-sided [-0.045 to 0.057], Standard Error of Mean 0.026 — spatial power covariance structure for within-patient errors

20. Secondary Outcome: Trough FVC Response on Day 170
Description: Trough FVC was defined as the FVC value at the end of the dosing interval (24 hours) and was calculated as the mean of the 2 FVC measurements performed at 23h and at 23h 50 min after inhalation of study medication at the clinic visit on the previous day.
  Trough FVC response was defined as trough FVC minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted means (SE) were obtained from fitting an MMRM including fixed effects of treatment, planned test day, treatment-by-test day interaction, baseline and baseline-by-test day interaction, patient as random effect, and spatial power covariance structure for within-patient errors and Kenward-Roger approximation for denominator degrees of freedom.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures (MMRM) model in each treatment group.
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and at 23h and at 23h 50 min after inhalation of study medication on day 170
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.116 (0.018) | 0.163 (0.018) | 0.202 (0.018) | 0.266 (0.018) | 0.274 (0.018)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.158, 95% CI 2-sided [0.108 to 0.208], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0048, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.072, 95% CI 2-sided [0.022 to 0.122], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.150, 95% CI 2-sided [0.101 to 0.200], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.103, 95% CI 2-sided [0.053 to 0.152], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0116, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.064, 95% CI 2-sided [0.014 to 0.113], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.7577, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.008, 95% CI 2-sided [-0.042 to 0.058], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.111, 95% CI 2-sided [0.061 to 0.160], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0007, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.086, 95% CI 2-sided [0.037 to 0.136], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0621, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.048, 95% CI 2-sided [-0.002 to 0.097], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1266, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.039, 95% CI 2-sided [-0.011 to 0.089], Standard Error of Mean 0.025 — spatial power covariance structure for within-patient errors

21. Secondary Outcome: Trough FVC Response on Day 365
Description: as for outcome 17
Time Frame: 1 h and 10 min prior to dose on the first day of randomized treatment (baseline) and on day 365
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 503 | 499 | 498 | 500 | 497
Litres | 0.028 (0.019) | 0.096 (0.019) | 0.097 (0.019) | 0.198 (0.019) | 0.184 (0.019)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.156, 95% CI 2-sided [0.104 to 0.209], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0013, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.087, 95% CI 2-sided [0.034 to 0.139], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.170, 95% CI 2-sided [0.118 to 0.223], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.102, 95% CI 2-sided [0.049 to 0.154], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.100, 95% CI 2-sided [0.048 to 0.153], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.6093, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.014, 95% CI 2-sided [-0.066 to 0.039], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.088, 95% CI 2-sided [0.035 to 0.140], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0095, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.070, 95% CI 2-sided [0.017 to 0.123], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0108, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.069, 95% CI 2-sided [0.016 to 0.121], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.9627, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.001, 95% CI 2-sided [-0.051 to 0.054], Standard Error of Mean 0.027 — spatial power covariance structure for within-patient errors

22. Secondary Outcome: FEV1 AUC(0-12h) Response in Sub-set of Patients With 12-hour Pulmonary Function Test (PFT) on Day 169 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: FEV1 AUC(0-12h) was calculated as the area under the FEV1- time curve from 0 to 12 h post-dose using the trapezoidal rule, divided by the duration (12 h) to report in litres.
  FEV1 AUC(0-12h) response was defined as FEV1 AUC(0-12h) minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted mean (SE) were obtained from fitting an ANCOVA model with categorical effect of treatment and baseline as covariate.
  Number of participants analyzed are the number of patients contributing to the ANCOVA model in each treatment group.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 169 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h post-dose on Day 169
Population: 12 hr PFT set: All patients who have given Informed Consent for the 12-hour PFT testing and had any spirometry measurement after 3-hour and before or at 12-hours post-dose on Days 169 and 170.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 194 | 185 | 160 | 178 | 167
Litres | 0.131 (0.015) | 0.109 (0.016) | 0.127 (0.017) | 0.202 (0.016) | 0.250 (0.016)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.118, 95% CI 2-sided [0.074 to 0.162], Standard Error of Mean 0.022
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.123, 95% CI 2-sided [0.077 to 0.169], Standard Error of Mean 0.023
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0012, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.071, 95% CI 2-sided [0.028 to 0.114], Standard Error of Mean 0.022
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.094, 95% CI 2-sided [0.050 to 0.137], Standard Error of Mean 0.022
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0010, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.076, 95% CI 2-sided [0.031 to 0.121], Standard Error of Mean 0.023
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0384, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.047, 95% CI 2-sided [0.003 to 0.092], Standard Error of Mean 0.023
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.141, 95% CI 2-sided [0.097 to 0.185], Standard Error of Mean 0.022
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8428, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.004, 95% CI 2-sided [-0.049 to 0.040], Standard Error of Mean 0.023
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.3048, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.022, 95% CI 2-sided [-0.065 to 0.020], Standard Error of Mean 0.022
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4311, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.018, 95% CI 2-sided [-0.027 to 0.063], Standard Error of Mean 0.023

23. Secondary Outcome: FEV1 AUC(0-24h) Response in Sub-set of Patients With 12-hour PFTs on Day 169 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: FEV1 AUC(0-24h) was calculated as the area under the FEV1- time curve from 0 to 24 h post-dose using the trapezoidal rule, divided by the duration (24 h) to report in litres. FEV1 AUC(0-24h) response was defined as FEV1 AUC(0-24h) minus baseline FEV1. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted mean (SE) were obtained from fitting an ANCOVA model with categorical effect of treatment and baseline as covariate.
  Number of participants analyzed are the number of patients contributing to the ANCOVA model in each treatment group.
Time Frame: 1 hour (h) and 10 minutes (min) prior to dose to on the first day of randomized treatment and on Day 169 and 5 min, 15 min, 30 min, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 8 h, 10 h, 12 h, 23 h, 23 h and 50 min post-dose on Day 169
Population: 12-hr PFT set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 194 | 185 | 160 | 178 | 167
Litres | 0.108 (0.014) | 0.083 (0.015) | 0.100 (0.016) | 0.159 (0.015) | 0.206 (0.015)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.098, 95% CI 2-sided [0.057 to 0.139], Standard Error of Mean 0.021
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.106, 95% CI 2-sided [0.063 to 0.149], Standard Error of Mean 0.022
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0136, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.051, 95% CI 2-sided [0.010 to 0.091], Standard Error of Mean 0.021
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0003, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.075, 95% CI 2-sided [0.035 to 0.116], Standard Error of Mean 0.021
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0065, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.059, 95% CI 2-sided [0.016 to 0.101], Standard Error of Mean 0.022
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0277, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.047, 95% CI 2-sided [0.005 to 0.089], Standard Error of Mean 0.021
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.122, 95% CI 2-sided [0.081 to 0.164], Standard Error of Mean 0.021
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.7116, ANCOVA — Comments ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.008, 95% CI 2-sided [-0.049 to 0.034], Standard Error of Mean 0.021
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.2332, ANCOVA — Comments ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.024, 95% CI 2-sided [-0.065 to 0.016], Standard Error of Mean 0.020
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.4374, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.017, 95% CI 2-sided [-0.025 to 0.059], Standard Error of Mean 0.021

24. Secondary Outcome: FVC AUC(0-12h) Response in Sub-set of Patients With 12-hour PFTs on Day 169 From Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: FVC AUC(0-12h) was calculated as the area under the FVC- time curve from 0 to 12 h post-dose using the trapezoidal rule, divided by the duration (12 h) to report in litres.
  FVC AUC(0-12h) response was defined as FVC AUC(0-12h) minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted mean (SE) were obtained from fitting an ANCOVA model with categorical effect of treatment and baseline as covariate. Number of participants analyzed are the number of patients contributing to the ANCOVA model in each treatment group.
Time Frame: as for outcome 22
Population: 12-hr PFT set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 194 | 185 | 160 | 178 | 167
Litres | 0.227 (0.029) | 0.180 (0.030) | 0.248 (0.032) | 0.356 (0.030) | 0.388 (0.031)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0002, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.161, 95% CI 2-sided [0.077 to 0.244], Standard Error of Mean 0.043
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0017, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.140, 95% CI 2-sided [0.053 to 0.228], Standard Error of Mean 0.045
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0022, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.128, 95% CI 2-sided [0.046 to 0.210], Standard Error of Mean 0.042
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.176, 95% CI 2-sided [0.093 to 0.259], Standard Error of Mean 0.042
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0141, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.108, 95% CI 2-sided [0.022 to 0.194], Standard Error of Mean 0.044
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4581, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.032, 95% CI 2-sided [-0.053 to 0.118], Standard Error of Mean 0.043
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.208, 95% CI 2-sided [0.124 to 0.293], Standard Error of Mean 0.043
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.6335, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.021, 95% CI 2-sided [-0.064 to 0.105], Standard Error of Mean 0.043
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.2530, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.047, 95% CI 2-sided [-0.129 to 0.034], Standard Error of Mean 0.041
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1188, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.068, 95% CI 2-sided [-0.017 to 0.153], Standard Error of Mean 0.043

25. Secondary Outcome: FVC AUC(0-24h) Response in Sub-set of Patients With 12-hour PFTs on Day 169 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: FVC AUC(0-24h) was calculated as the area under the FVC- time curve from 0 to 24 h post-dose using the trapezoidal rule, divided by the duration (24 h) to report in litres.
  FVC AUC(0-24h) response was defined as FVC AUC(0-24h) minus baseline FVC. Baseline was defined as the mean of the 2 pre-dose measurements performed 1 h and 10 min prior to administration of the first dose at visit 2 (day 1).
  The adjusted mean (SE) were obtained from fitting an ANCOVA model with categorical effect of treatment and baseline as covariate.
  Number of participants analyzed are the number of patients contributing to the ANCOVA model in each treatment group.
Time Frame: as for outcome 23
Population: 12-hr PFT set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 194 | 185 | 160 | 178 | 167
Litres | 0.192 (0.028) | 0.141 (0.028) | 0.203 (0.030) | 0.297 (0.029) | 0.329 (0.030)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0008, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.137, 95% CI 2-sided [0.057 to 0.217], Standard Error of Mean 0.041
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0032, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.126, 95% CI 2-sided [0.042 to 0.209], Standard Error of Mean 0.043
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0085, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.105, 95% CI 2-sided [0.027 to 0.183], Standard Error of Mean 0.040
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.156, 95% CI 2-sided [0.077 to 0.235], Standard Error of Mean 0.040
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0255, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.094, 95% CI 2-sided [0.011 to 0.176], Standard Error of Mean 0.042
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4393, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.032, 95% CI 2-sided [-0.049 to 0.113], Standard Error of Mean 0.041
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.188, 95% CI 2-sided [0.108 to 0.269], Standard Error of Mean 0.041
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.7784, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.012, 95% CI 2-sided [-0.069 to 0.092], Standard Error of Mean 0.041
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1965, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = -0.051, 95% CI 2-sided [-0.129 to 0.026], Standard Error of Mean 0.039
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1315, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Adjusted mean difference = 0.063, 95% CI 2-sided [-0.019 to 0.144], Standard Error of Mean 0.041

26. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score on Day 85 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: as for outcome 3
Time Frame: Day 85
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 954 | 960 | 955 | 990 | 979
points on a scale | 38.832 (0.398) | 37.821 (0.397) | 37.822 (0.399) | 37.304 (0.392) | 36.691 (0.394)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -2.141, 95% CI 2-sided [-3.239 to -1.043], Standard Error of Mean 0.560 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0435, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.131, 95% CI 2-sided [-2.230 to -0.033], Standard Error of Mean 0.560 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0063, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.528, 95% CI 2-sided [-2.623 to -0.432], Standard Error of Mean 0.559 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.3545, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.517, 95% CI 2-sided [-1.611 to 0.577], Standard Error of Mean 0.558 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.3542, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.518, 95% CI 2-sided [-1.614 to 0.578], Standard Error of Mean 0.559 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2697, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.613, 95% CI 2-sided [-1.702 to 0.476], Standard Error of Mean 0.556 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0434, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.130, 95% CI 2-sided [-2.227 to -0.033], Standard Error of Mean 0.559 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0732, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.010, 95% CI 2-sided [-2.114 to 0.095], Standard Error of Mean 0.563 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0724, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.011, 95% CI 2-sided [-2.114 to 0.092], Standard Error of Mean 0.563 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.9983, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.001, 95% CI 2-sided [-1.102 to 1.104], Standard Error of Mean 0.563 — Spatial power covariance structure for within-patient errors

27. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score on Day 365 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: as for outcome 3
Time Frame: Day 365
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 954 | 960 | 955 | 990 | 979
points on a scale | 38.989 (0.414) | 37.609 (0.409) | 37.581 (0.411) | 37.553 (0.403) | 37.138 (0.404)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.852, 95% CI 2-sided [-2.985 to -0.718], Standard Error of Mean 0.578 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4413, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.444, 95% CI 2-sided [-1.573 to 0.686], Standard Error of Mean 0.576 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0129, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.437, 95% CI 2-sided [-2.569 to -0.304], Standard Error of Mean 0.578 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.9222, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.056, 95% CI 2-sided [-1.182 to 1.070], Standard Error of Mean 0.574 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.9602, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.029, 95% CI 2-sided [-1.157 to 1.100], Standard Error of Mean 0.576 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4669, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.415, 95% CI 2-sided [-1.533 to 0.703], Standard Error of Mean 0.570 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.4126, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.471, 95% CI 2-sided [-1.598 to 0.656], Standard Error of Mean 0.575 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0158, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.408, 95% CI 2-sided [-2.551 to -0.265], Standard Error of Mean 0.583 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.0177, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -1.381, 95% CI 2-sided [-2.521 to -0.240], Standard Error of Mean 0.582 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.9624, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.027, 95% CI 2-sided [-1.164 to 1.109], Standard Error of Mean 0.580 — Spatial power covariance structure for within-patient errors

28. Secondary Outcome: Mahler Transitional Dyspnoea Index (TDI) Focal Score on Day 43 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: Mahler TDI focal score on Day 43 From the two twin trials, present 1237.6 (NCT01431287) and 1237.5 (NCT01431274).
  The Mahler Dyspnoea questionnaire is an instrument which measures change from the baseline state The TDI focal score was used to measure the effect of Tio+Olo FDC on patients' dyspnoea after 24 weeks of treatment (Day 169). The focal score is the sum of the subscale scores for Functional Impairment, Magnitude of Effort and Magnitude of Task. Scores for each subscale range from -3 to 3 so that the Focal score ranges from -9 to 9. For all subscale scores and the Focal score a higher value indicates a better outcome.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 43
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 984 | 982 | 978 | 992 | 992
points on a scale | 1.453 (0.096) | 1.430 (0.097) | 1.408 (0.097) | 1.876 (0.096) | 2.048 (0.096)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.595, 95% CI 2-sided [0.329 to 0.862], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.640, 95% CI 2-sided [0.373 to 0.907], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0019, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.423, 95% CI 2-sided [0.156 to 0.690], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0011, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.446, 95% CI 2-sided [0.179 to 0.712], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0006, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.468, 95% CI 2-sided [0.201 to 0.735], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.2045, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.172, 95% CI 2-sided [-0.094 to 0.438], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.618, 95% CI 2-sided [0.351 to 0.885], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.7432, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.045, 95% CI 2-sided [-0.313 to 0.223], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.8687, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.023, 95% CI 2-sided [-0.290 to 0.245], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.8709, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = -0.022, 95% CI 2-sided [-0.290 to 0.246], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors

29. Secondary Outcome: Mahler Transitional Dyspnoea Index (TDI) Focal Score on Day 85 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: Mahler TDI focal score on Day 85 From the two twin trials, present 1237.6 (NCT01431287) and 1237.5 (NCT01431274).
  The Mahler Dyspnoea questionnaire is an instrument which measures change from the baseline state The TDI focal score was used to measure the effect of Tio+Olo FDC on patients' dyspnoea after 24 weeks of treatment (Day 169). The focal score is the sum of the subscale scores for Functional Impairment, Magnitude of Effort and Magnitude of Task. Scores for each subscale range from -3 to 3 so that the Focal score ranges from -9 to 9. For all subscale scores and the Focal score a higher value indicates a better outcome.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 85
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 984 | 982 | 978 | 992 | 992
points on a scale | 1.506 (0.097) | 1.698 (0.097) | 1.702 (0.097) | 1.925 (0.096) | 2.136 (0.096)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.630, 95% CI 2-sided [0.362 to 0.898], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0015, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.434, 95% CI 2-sided [0.166 to 0.703], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0022, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.419, 95% CI 2-sided [0.151 to 0.687], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0966, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.227, 95% CI 2-sided [-0.041 to 0.495], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.1029, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.223, 95% CI 2-sided [-0.045 to 0.492], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.1220, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.211, 95% CI 2-sided [-0.056 to 0.478], Standard Error of Mean 0.136 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.438, 95% CI 2-sided [0.170 to 0.707], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.1542, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.196, 95% CI 2-sided [-0.074 to 0.465], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.1626, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.192, 95% CI 2-sided [-0.077 to 0.461], Standard Error of Mean 0.137 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.9765, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; djusted mean difference = 0.004, 95% CI 2-sided [-0.265 to 0.274], Standard Error of Mean 0.138 — Spatial power covariance structure for within-patient errors

30. Secondary Outcome: Mahler Transitional Dyspnoea Index (TDI) Focal Score on Day 365 From the Two Twin Trials, Present 1237.6 (NCT01431287) and 1237.5 (NCT01431274)
Description: Mahler TDI focal score on Day 365 From the two twin trials, present 1237.6 (NCT01431287) and 1237.5 (NCT01431274).
  The Mahler Dyspnoea questionnaire is an instrument which measures change from the baseline state The TDI focal score was used to measure the effect of Tio+Olo FDC on patients' dyspnoea after 24 weeks of treatment (Day 169). The focal score is the sum of the subscale scores for Functional Impairment, Magnitude of Effort and Magnitude of Task. Scores for each subscale range from -3 to 3 so that the Focal score ranges from -9 to 9. For all subscale scores and the Focal score a higher value indicates a better outcome.
  Number of participants analyzed are the number of patients contributing to the mixed effect repeated measures model (MMRM) in each treatment group.
Time Frame: Day 365
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: points on a scale
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Number analyzed (Participants) | 984 | 982 | 978 | 992 | 992
points on a scale | 1.411 (0.101) | 1.450 (0.100) | 1.736 (0.101) | 1.782 (0.099) | 2.058 (0.099)
Statistical Analysis 1: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.647, 95% CI 2-sided [0.370 to 0.925], Standard Error of Mean 0.142 — Spatial power covariance structure for within-patient errors
Statistical Analysis 2: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0226, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.322, 95% CI 2-sided [0.045 to 0.600], Standard Error of Mean 0.141 — Spatial power covariance structure for within-patient errors
Statistical Analysis 3: Comparison: Olodaterol (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0089, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.371, 95% CI 2-sided [0.093 to 0.649], Standard Error of Mean 0.142 — Spatial power covariance structure for within-patient errors
Statistical Analysis 4: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.0186, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.332, 95% CI 2-sided [0.056 to 0.609], Standard Error of Mean 0.141 — Spatial power covariance structure for within-patient errors
Statistical Analysis 5: Comparison: Tiotropium (5 μg) vs Tio+Olo FDC (2.5/5 μg); Test type: Superiority or Other; p = 0.7441, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.046, 95% CI 2-sided [-0.231 to 0.324], Standard Error of Mean 0.142 — Spatial power covariance structure for within-patient errors
Statistical Analysis 6: Comparison: Tio+Olo FDC (2.5/5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p = 0.0492, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.276, 95% CI 2-sided [0.001 to 0.551], Standard Error of Mean 0.140 — Spatial power covariance structure for within-patient errors
Statistical Analysis 7: Comparison: Tiotropium (2.5 μg) vs Tio+Olo FDC (5/5 μg); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.608, 95% CI 2-sided [0.332 to 0.884], Standard Error of Mean 0.141 — Spatial power covariance structure for within-patient errors
Statistical Analysis 8: Comparison: Olodaterol (5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0230, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.325, 95% CI 2-sided [0.045 to 0.605], Standard Error of Mean 0.143 — Spatial power covariance structure for within-patient errors
Statistical Analysis 9: Comparison: Olodaterol (5 μg) vs Tiotropium (2.5 μg); Test type: Superiority or Other; p = 0.7855, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.039, 95% CI 2-sided [-0.240 to 0.317], Standard Error of Mean 0.142 — Spatial power covariance structure for within-patient errors
Statistical Analysis 10: Comparison: Tiotropium (2.5 μg) vs Tiotropium (5 μg); Test type: Superiority or Other; p = 0.0442, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Kenward-Roger approximation of denominator degrees of freedom; Adjusted mean difference = 0.286, 95% CI 2-sided [0.007 to 0.564], Standard Error of Mean 0.142 — Spatial power covariance structure for within-patient errors

ADVERSE EVENTS:
Time Frame: All Adverse events with an onset after the first dose of study medication up to a period of 21 days after the last dose of study medication were assigned to the treatment period for evaluation (Up to 459 days)
Groups:
- Olodaterol (5 μg): Oral inhalation of Olodaterol 5 μg (2.5 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tiotropium (2.5 μg): Oral inhalation of Tiotropium 2.5 μg (1.25 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tiotropium (5 μg): Oral inhalation of Tiotropium 5 μg (2.5 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tio+Olo FDC (2.5/5 μg): Oral inhalation of fixed dose combination (FDC) of Tiotropium 2.5 μg and Olodaterol 5 μg (Tiotropium: 1.25 μg per actuation and Olodaterol: 2.5 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
- Tio+Olo FDC (5/5 μg): Oral inhalation of FDC of Tiotropium 5 μg and Olodaterol 5 μg (Tiotropium and Olodaterol: 2.5 μg per actuation) , 2 puffs from the RESPIMAT inhaler, once daily, in the morning.
Arm/Group | Olodaterol (5 μg) | Tiotropium (2.5 μg) | Tiotropium (5 μg) | Tio+Olo FDC (2.5/5 μg) | Tio+Olo FDC (5/5 μg)
Serious Adverse Events (participants affected / at risk) | 106/510 | 90/507 | 93/506 | 87/508 | 82/507
Other Adverse Events (participants affected / at risk) | 246/510 | 228/507 | 216/506 | 223/508 | 214/507
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5 μg) (N=510) | Tiotropium (2.5 μg) (N=507) | Tiotropium (5 μg) (N=506) | Tio+Olo FDC (2.5/5 μg) (N=508) | Tio+Olo FDC (5/5 μg) (N=507)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 3 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 2 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0 | 2 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 1 | 3 | 1 | 2
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Malformation biliary (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0
Age-related macular degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0
Macular degeneration (Eye disorders) | 0 | 1 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 1 | 2 | 0
Death (General disorders) | 1 | 1 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 0 | 0 | 1 | 1
Drowning (General disorders) | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Medical device complication (General disorders) | 0 | 1 | 0 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 2
Bronchopneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 1 | 0 | 1
Cellulitis pharyngeal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Dermatitis infected (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Graft infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 1 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 6 | 6 | 2 | 9 | 9
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Superinfection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 2 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Liver contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Troponin T increased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Bone deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 2 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Sweat gland tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Acute polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 2 | 0 | 2
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neuromyopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 1 | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1
Renal vasculitis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 4 | 1 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2 | 0
Analgesic asthma syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 41 | 37 | 33 | 30 | 33
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 3 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 3
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Arteritis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Leriche syndrome (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Shock (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olodaterol (5 μg) (N=510) | Tiotropium (2.5 μg) (N=507) | Tiotropium (5 μg) (N=506) | Tio+Olo FDC (2.5/5 μg) (N=508) | Tio+Olo FDC (5/5 μg) (N=507)
Nasopharyngitis (Infections and infestations) | 66 | 59 | 54 | 70 | 61
Upper respiratory tract infection (Infections and infestations) | 32 | 31 | 27 | 29 | 29
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 147 | 146 | 132 | 118 | 129
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 27 | 25 | 29 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 22 | 27 | 21 | 20
Hypertension (Vascular disorders) | 26 | 10 | 10 | 19 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.